CLINICAL TRIAL: NCT00864786
Title: A Double Blind (3rd Party Open), Randomised, Placebo Controlled, Dose Escalating Study To Investigate The Safety, Toleration, Pharmacokinetics, And Pharmacodynamics Of Multiple Inhaled Doses Of PF-03635659 In Healthy Male Subjects.
Brief Title: Multiple Dose Healthy Volunteer Safety Pharmacokinetics Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B0431002
Record Dates: First submitted 2008-12-22; First posted 2009-03-19 (Estimated); Last update posted 2009-03-23 (Estimated); Status verified 2009-03

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Multiple dose safety and pharmacokinetics study
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (5):
- Cohort 1 (Experimental): 200 mcg
  Interventions: Drug: PF03635659
- Cohort 2 (Experimental): 600 mcg
  Interventions: Drug: PF03635659
- Cohort 3 (Experimental): 1000 mcg
  Interventions: Drug: PF03635659
- Cohort 4 (Experimental): Dose to be decided
  Interventions: Drug: PF03635659
- Cohort 5 (Experimental): Dose to be decided
  Interventions: Drug: PF03635659

INTERVENTIONS:
Drug: PF03635659 — Inhaled doses of 200 mcgQD
  Arms: Cohort 1
Drug: PF03635659 — Inhaled doses of 600 mcg QD
  Arms: Cohort 2
Drug: PF03635659 — Inhaled doses of 1000 mcg QD
  Arms: Cohort 3
Drug: PF03635659 — Inhaled dose to be decided based on all available data from previous cohorts. It will run if maximum tolerated dose is not identified from previous cohorts or if a lower dose is required to be investigated.
  Arms: Cohort 4
Drug: PF03635659 — Inhaled dose to be decided based on all available data from previous cohorts. It will run if maximum tolerated dose is not identified from previous cohorts or if a lower dose is required to be investigated.
  Arms: Cohort 5

SUMMARY:
Multiple dose safety and pharmacokinetics in healthy male subjects

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects between the ages of 18 and 55 years, inclusive (Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12-lead ECG and clinical laboratory tests).
* Body Mass Index (BMI) of approximately 18 to 30 kg/m2; and a total body weight >50 kg (110 lbs). A BMI lower limit of 17.5 kg/m2 may be rounded up to 18.0 kg/m2; a BMI upper limit of 30.5 kg/m2 may be rounded down to 30.0 kg/m2 and will be acceptable for inclusion.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing) disease or clinical findings at screening.
* Any condition possibly affecting drug absorption (eg, gastrectomy).

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2008-09; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Safety and toleration: Adverse events, vital signs measurements (supine and standing), 12-lead ECGs, spirometry (FEV1, FVC), laboratory safety tests, physical examination, and subject-reported dry mouth assessment. | 3 Weeks
Pharmacokinetics: Plasma: Cmax, Tmax, AUCinf, AUCτ, t½, accumulation ratio, linearity ratio. | 3 Weeks
Pharmacodynamics: Salivary flow rate | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Brussels, Belgium

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B0431002&StudyName=Multiple%20dose%20healthy%20volunteer%20safety%20pharmacokinetics%20study